CLINICAL TRIAL: NCT06221540
Title: The Impact of an Evidence-based Myth-busting Information Intervention on Maternal Food Allergy Related Quality of Life, Anxiety and Self-efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Health Ireland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GEN/894/21
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Child Allergy; Food Allergy
Keywords: Educational intervention; Food Allergy; Quality of Life; Anxiety; Self efficacy; Maternal education; Booklet; Immune System Diseases; Hypersensitivity, Immediate; Food Hypersensitivity
MeSH Terms: conditions — Food Hypersensitivity; Anxiety Disorders; Immune System Diseases; Hypersensitivity, Immediate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Received written patient information leaflet (Experimental)
  Interventions: Behavioral: "Myth busting" information leaflet
- Routine education at first clinic appointment (No Intervention): Active Comparator

INTERVENTIONS:
Behavioral: "Myth busting" information leaflet — A written patient information leaflet displaying ten food allergy myths with the myth-busting evidence-based information clearly stated, focusing on themes pertinent to the myth-busting information
  Arms: Received written patient information leaflet

SUMMARY:
Children with Food Allergy (FA) are at risk of life threatening reactions. They must carry an emergency medicine kit containing adrenaline auto-injector devices for the immediate treatment of anaphylaxis.

Much research has documented the adverse impact of childhood FA on the food allergy related quality of life (FQoL) of the Carer and the family, along with reported higher levels of anxiety and stress. These adverse impacts are largely driven by the need for Carers to always be "emergency ready". Mothers of food allergic children report higher levels of anxiety compared to the rest of the family, possibly due to mothers commonly being the primary care givers responsible for the preparation of meals, childcare etc.

Carers of newly diagnosed food allergic children, looking for more information about their child's FA are at risk of exposure to myths and misinformation about food allergy. These falsehoods are likely to increase further, Carers Food Allergy-related anxiety.

The investigators wish to survey the frequency with which common myths on FA are believed among mothers prior to their attendance at an allergy clinic. They wish to understand the impact of "myth-busting" information on maternal anxiety or self-efficacy when provided to mothers while awaiting a specialist appointment.

The research question is to determine if the online educational session is effective at decreasing anxiety and improving quality of life in Carers of FA children awaiting a specialist appointment.

DETAILED DESCRIPTION:
Carers of food allergic children report that their information needs are greatest at the beginning of their journey when their child first experiences a food allergic reaction. Unfortunately, wait times to attend specialist paediatric allergy clinics can be lengthy. Thus, families can experience a prolonged time-gap between the initial allergic reaction and accessing diagnostic testing and benefitting from multi-disciplinary support and education. Furthermore, carers report often contradictory advice from non-specialist Healthcare Professionals (HCPs). This in turn encourages carers to look for information online with many using search engines unless guided to official food allergy websites by HCPs. Not all online information is correct, or evidence based. Often information provided suggests that certain FA children are at greater risk of anaphylaxis and mortality. This in turn increases anxiety amongst carers and impairs their quality of life.

The purpose of this study is to develop an effective intervention that improves maternal FA related quality of life, anxiety, and self-efficacy prior to attending their child's first paediatric allergy clinic appointment. A randomized control trial will be performed comparing quality of life, anxiety and self efficacy in carers who receive the intervention versus those that do not. Participants will be randomized into 2 groups. All volunteers, from both groups, will complete questionnaires online using only a study identifier number. This will ensure anonymity throughout the study. The only personal information that will be asked is the carer's age group, whether they are a mother or father, their child's age and gender and whether they have any other allergies. Group 1 will be sent a written patient information leaflet displaying ten food allergy myths with the myth-busting evidence-based information clearly stated. Two weeks following the online educational session, Groups 1 and 2 will again complete the online questionnaires.

The outcomes are health related quality of life and levels of anxiety. It is hoped that the findings will positively support Carers, children and their families

ELIGIBILITY:
Inclusion Criteria:

* First referral to Children's Health Ireland allergy service for evaluation of 'Immediate type' IgE food allergy.
* Referral accepted and triaged to a waiting list between 30 months to six months prior to study commencement.
* Child aged between three years and 12 years at the time of study commencement.

Exclusion Criteria:

* Referral source from Children's Health Ireland (CHI) dermatology or immunology services or the patient already attends services that will evaluate food allergy such as CHI dermatology and /or immunology.
* Child younger than three years and older than 12 years at the time of study commencement.
* Referral information is not suggestive of an IgE mediated food allergy.
* Complex referral history suggestive of chronic urticaria, mast cell disorders or eosinophilic oesophagitis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Primary Outcome 1 | 2 weeks
  Change in score in each group on Food Allergy Quality of Life Questionnaire (FAQLQ)-Parental Proxy Form
Primary Outcome 2 | 2 weeks
  Change in score in each group on Food Allergy Independent Measurement (FAIM)
Primary Outcome 3 | 2 weeks
  Change in score in each group on Food Allergy Anxiety Scale (FAAS)

SECONDARY OUTCOMES:
Secondary score | 2 weeks
  Agreement with Food Allergy Myths measured using the Food Allergy Belief (FAB) scale (SEFAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Aideen Byrne, PhD, Principal Investigator — Children's Health Ireland
Locations (1):
- Children's Health Ireland, Dublin, Ireland